CLINICAL TRIAL: NCT01022788
Title: Improving Newborn Survival in Rural Southern Tanzania: a Study to Evaluate the Impact and Cost of a Scaleable Package of Interventions at Community Level With Health System Strengthening
Brief Title: Improving Newborn Survival In Southern Tanzania
Acronym: INSIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Save the Children (Other); UNICEF (Other)
Responsible Party: Principal Investigator, Joanna Schellenberg, Professor of Epidemiology and International Health, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5316
Record Dates: First submitted 2009-11-27; First posted 2009-12-01 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Newborn Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home-based counselling visits by volunteers (Experimental): Home-based counselling in pregnancy and the first few days of life to encourage women and families to adopt key newborn care behaviours
  Interventions: Behavioral: Home-based counselling
- Standard care through existing health system (No Intervention)

INTERVENTIONS:
Behavioral: Home-based counselling
  Other Names: Mtunze Mtoto Mchanga
  Arms: Home-based counselling visits by volunteers

SUMMARY:
This study will develop, implement and evaluate the effectiveness and cost of interventions at community level (focussed on a community-based health worker) and of health system strengthening on newborn survival in rural southern Tanzania.

Objectives

1. To develop and document a community-based package for improved newborn care, focussed around interpersonal communication through home visits in pregnancy and the early neonatal period .
2. To develop and document a quality improvement package for antenatal, intrapartum and postnatal care in health facilities.
3. To implement these strategies for improved newborn survival in such a way as to be both sustainable and scaleable at national level.
4. To monitor understanding of, and attitudes related to, neonatal care and survival from both health provider and community perspectives in areas with and without the interventions.
5. To measure incremental costs and cost savings to the health sector and society associated with the interventions, and to predict the cost of integrating the programme into routine health service provision and of scaling-up
6. To strengthen Tanzania's capacity to develop, implement and evaluate interventions to improve neonatal survival.
7. To estimate the effect of the interventions on newborn survival and household behaviours related to newborn health.

Study design & methods. The interventions will be implemented in parts of Lindi and Mtwara regions. The health system quality improvement package will be implemented throughout the area and evaluated using a before-after comparison. The community intervention will be implemented initially in a randomly-chosen half of all wards (a ward is an administrative sub-area of a district). Implementation will be led by existing front-line health staff. Evaluation will include a health facility survey and a household survey to assess contacts with the agents of change, key behaviours and newborn survival in the community.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women living in the study area

Exclusion Criteria:

* Unwilling to participate

Max Age: 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 47688 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Newborn survival (to 28 days) | July 2010 to June 2013

SECONDARY OUTCOMES:
Household behaviours for essential newborn care | July 2010 to June 2013

CONTACTS AND LOCATIONS:
Overall Officials: David Schellenberg, Principal Investigator — London School of Hygiene and Tropical Medicine; Hassan Mshinda, Principal Investigator — Ifakara Health Institute and COSTECH; Marcel Tanner, Principal Investigator — Swiss Tropical & Public Health Institute; Fatuma Manzi, PhD, Principal Investigator — Ifakara Health Institute, Tanzania
Locations (1):
- Mtwara R, Tandahimba, Newala, Nachingwea, Lindi R, Ruangwa, Mtwara and Lindi Regions, Tanzania

REFERENCES:
- [Derived] Hanson C, Manzi F, Mkumbo E, Shirima K, Penfold S, Hill Z, Shamba D, Jaribu J, Hamisi Y, Soremekun S, Cousens S, Marchant T, Mshinda H, Schellenberg D, Tanner M, Schellenberg J. Effectiveness of a Home-Based Counselling Strategy on Neonatal Care and Survival: A Cluster-Randomised Trial in Six Districts of Rural Southern Tanzania. PLoS Med. 2015 Sep 29;12(9):e1001881. doi: 10.1371/journal.pmed.1001881. eCollection 2015 Sep. PMID 26418813
- [Derived] Penfold S, Manzi F, Mkumbo E, Temu S, Jaribu J, Shamba DD, Mshinda H, Cousens S, Marchant T, Tanner M, Schellenberg D, Schellenberg JA. Effect of home-based counselling on newborn care practices in southern Tanzania one year after implementation: a cluster-randomised controlled trial. BMC Pediatr. 2014 Jul 22;14:187. doi: 10.1186/1471-2431-14-187. PMID 25052850
- [Derived] Mkumbo E, Hanson C, Penfold S, Manzi F, Schellenberg J. Innovation in supervision and support of community health workers for better newborn survival in southern Tanzania. Int Health. 2014 Dec;6(4):339-41. doi: 10.1093/inthealth/ihu016. Epub 2014 Apr 7. PMID 24711599